CLINICAL TRIAL: NCT03441724
Title: Mechanocardiographic Detection of Acute ST-Segment Elevation Myocardial Infarction - the MECHANO-STEMI Study
Brief Title: Mechanocardiography in Patients With STEMI
Acronym: MECHANO-STEMI
Status: Active, not recruiting | Type: Observational
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Juhani Airaksinen, Professor, University of Turku
Other Study IDs: T02/006/15
Record Dates: First submitted 2018-02-07; First posted 2018-02-22 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Myocardial Infarction, Acute
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- STEMI before PCI: ST-segment elevation, recording acquired before coronary intervention
  Interventions: Diagnostic Test: Mechanocardiography
- STEMI after PCI: ST-segment elevation, recording acquired from the same patients after coronary intervention
  Interventions: Diagnostic Test: Mechanocardiography

INTERVENTIONS:
Diagnostic Test: Mechanocardiography — Mechanocardiographic recording

SUMMARY:
The study aim is to evaluate the capability of mechanocardiography in detecting acute myocardial ischemia in patients suffering evolving ST-segment elevation infarction.

DETAILED DESCRIPTION:
Subsequent patients with ST-segment elevation assigned to the Turku University Hospital Heart Center cathlab for primary percutaneous coronary intervention are enrolled in the study. A 2 to 15 minutes mechanocardiographic recording is acquired before the intervention. A control recording is collected after the coronary intervention, within 24 hours. These recordings are compared and the results analyzed to determine the ability of this novel modality to discriminate between the two circumstances.

ELIGIBILITY:
Inclusion Criteria:

* Myocardial ischemia with ST-segment elevation in ECG
* Primary PCI procedure

Exclusion Criteria:

* Age >17 years
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Consecutive patients presenting with ST-segment elevation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Observed difference in mechanocardiographic signal | 24 hours
  In this novel method for recording cardiac mechanics, we anticipate to observe a difference in machanocardiography signal between the two states - before and after an occlusion of a coronary artery. As of yet, the precise nature of the signal change is unclear and will be clarified as the recorded signals are analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided